CLINICAL TRIAL: NCT01453855
Title: A Multicenter, Double-Masked Study of the Safety and Efficacy of Travoprost Ophthalmic Solution, 0.003% Compared to TRAVATAN in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Travoprost 3-Month Safety and Efficacy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-11-034; 2011-004587-29 (EudraCT Number)
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost 0.003% (Experimental): Travoprost ophthalmic solution, 0.003%, one drop instilled in each eye, once daily, for three months
  Interventions: Drug: Travoprost ophthalmic solution, 0.003%
- TRAVATAN (Active Comparator): Travoprost ophthalmic solution, 0.004%, one drop instilled in each eye, once daily, for three months
  Interventions: Drug: Travoprost ophthalmic solution, 0.004%

INTERVENTIONS:
Drug: Travoprost ophthalmic solution, 0.003%
  Arms: Travoprost 0.003%
Drug: Travoprost ophthalmic solution, 0.004%
  Other Names: TRAVATAN®
  Arms: TRAVATAN

SUMMARY:
The purpose of this study was to demonstrate that the intraocular pressure-lowering efficacy of Travoprost 0.003% is equivalent to TRAVATAN® in adult patients with open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This study consisted of six visits conducted during two sequential phases. The Screening/Eligibility phase included one screening visit and two eligibility visits. A washout period based on previous ocular medication preceded Eligibility Visit 1. Subjects who met all inclusion/exclusion criteria at both eligibility visits were randomized (1:1) at the second eligibility visit. The Treatment phase consisted of three on-therapy visits (Week 2, Week 6, and Month 3).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma (including open-angle glaucoma with pseudoexfoliation or pigment dispersion) or ocular hypertension.
* Qualifying intraocular pressure at both eligibility visits.
* Understand and sign an informed consent form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential if pregnant, breast-feeding, or not on adequate birth control.
* Severe central visual field loss in either eye.
* Chronic, recurrent or severe inflammatory eye disease.
* Best corrected visual acuity (BCVA) score worse than 55 ETDRS letters (equivalent to 20/80 Snellen).
* Any abnormality preventing reliable applanation tonometry.
* Hypersensitivity to prostaglandin analogs or to any component of the study medications.
* Therapy with another investigational agent within 30 days prior to the Screening Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1099 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Landry, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 60 investigational centers, including 52 in the US, 2 each in Sweden, Germany, and Austria, and 1 each in Spain and Finland.
Pre-assignment Details: Of the 1099 enrolled, 235 did not meet inclusion/exclusion criteria and were exited from the study prior to randomization. This reporting group includes all randomized subjects (864).
Period: Overall Study
Arm/Group | Travoprost 0.003% | TRAVATAN
Started | 442 | 422
Completed | 432 | 408
Not Completed | 10 | 14
Not completed — Adverse Event | 3 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Patient Decision Unrel to Adverse Event | 3 | 3
Not completed — Noncompliance | 1 | 0
Not completed — Inadequate Control of IOP | 1 | 5
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes subjects exposed to the study medication. Note: One subject in the TRAVATAN arm was randomized but discontinued prior to exposure to study medication and is not included in this reporting group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost 0.003% | TRAVATAN | Total
Number analyzed (Participants) | 442 | 421 | 863
Age, Customized [Number; unit: Participants]
  18 to 64 years | 189 | 193 | 382
  ≥ 65 years | 253 | 228 | 481
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 246 | 515
  Male | 173 | 175 | 348

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP) at Week 2, Week 6, and Month 3 for Each Assessment Time Point (8 AM, 10 AM, and 4 PM)
Description: As measured by Goldmann applanation tonometry. One eye from each subject was chosen as the study eye and only the study eye was used in the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Week 2, Week 6, Month 3 (8 AM, 10 AM, 4 PM)
Population: The intent-to-treat (ITT) analysis set included all patients who received study drug and completed at least 1 scheduled on-therapy study visit. In addition, no imputation methods were employed; therefore only efficacy measurements available at each visit and time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: millimeters mercury (mmHg)
Arm/Group | Travoprost 0.003% | TRAVATAN
Number analyzed (Participants) | 442 | 416
millimeters mercury (mmHg)
  Week 2 at 8 AM | 19.4 (0.16) | 19.5 (0.17)
  Week 2 at 10 AM | 18.6 (0.16) | 18.6 (0.16)
  Week 2 at 4 PM | 18.0 (0.16) | 18.3 (0.16)
  Week 6 at 8 AM | 19.3 (0.16) | 19.3 (0.17)
  Week 6 at 10 AM | 18.5 (0.16) | 18.6 (0.17)
  Week 6 at 4 PM | 18.0 (0.16) | 18.1 (0.17)
  Month 3 at 8 AM | 19.2 (0.17) | 19.3 (0.18)
  Month 3 at 10 AM | 18.3 (0.17) | 18.6 (0.18)
  Month 3 at 4 PM | 18.0 (0.16) | 18.0 (0.17)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment to study completion. An adverse event was considered to be any untoward medical occurrence in a patient exposed to the study medication.
Description: This reporting group includes subjects exposed to the study medication.
Arm/Group | Travoprost 0.003% | TRAVATAN
Serious Adverse Events (participants affected / at risk) | 5/442 | 7/421
Other Adverse Events (participants affected / at risk) | 56/442 | 64/421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travoprost 0.003% (N=442) | TRAVATAN (N=421)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 2 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Travoprost 0.003% (N=442) | TRAVATAN (N=421)
Ocular hyperaemia (Eye disorders) | 31 | 34
Conjunctival hyperaemia (Eye disorders) | 25 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.